CLINICAL TRIAL: NCT00237406
Title: Interactive Voice Response for Methadone Patients
Brief Title: Interactive Voice Response (IVR) for Methadone Patients
Status: Completed | Type: Observational
Sponsor: Butler Hospital (Other)
Other Study IDs: 4065-05
Record Dates: First submitted 2005-10-11; First posted 2005-10-12 (Estimated); Last update posted 2010-03-25 (Estimated); Status verified 2010-03

CONDITIONS: Opioid-Related Disorders
Keywords: IVR, methadone; methadone maintenance
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Procedure: interactive voice response

SUMMARY:
This study is designed to test whether a telephone call-in program is a feasible way to collect mood and drug-related information in individuals enrolled in a methadone maintenance program.

DETAILED DESCRIPTION:
Participants will complete a baseline interview and a follow-up interview at 5-weeks post-baseline. Two-thirds of the participants will be randomized into the telephone call-in group, and will be asked to complete daily, 10-minute, telephone interviews. To complete these interviews, participants will call into a toll-free telephone interview system with a unique and private Study ID number, and answers questions by using the telephone key pad. Questions during both the face-to-face interviews and the telephone interviews will assess mood, sleep, treatment utilization and drug-related experiences. Participants will be compensated for their time.

Comparison(s): Participants randomized into the telephone component of the study as compared to participants in the interview-only component of the study.

ELIGIBILITY:
Inclusion Criteria:

* Recent enrollment in a methadone maintenance program

Exclusion Criteria:

* Enrollment in a methadone maintenance program within the prior 3 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who recently enrolled in methadone maintenance for opioid addiction.
Sampling Method: Probability Sample
Enrollment: 50
Dates: Start 2006-01; Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Stein, MD, Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States